CLINICAL TRIAL: NCT00264875
Title: An Open-Label, Extension Safety And Efficacy Trial Of Pregabalin In Subjects With Neuropathic Pain Associated With Human Immunodeficiency Virus (HIV) Neuropathy
Brief Title: Open Label Safety And Efficacy Study Of Pregabalin In Subjects With Nerve Pain Asociated With Human Immunodeficiency Virus (HIV) Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081095
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Results first posted 2009-03-23 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Neuropathy; HIV Infections
MeSH Terms: conditions — Peripheral Nervous System Diseases; HIV Infections | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — 75mg BID, titrated up to 300mg according to individual response and tolerability

SUMMARY:
To evaluate the safety and efficacy of pregabalin in reducing neuropathic pain associated with HIV neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Participation in the preceding A0081066 double-blind trial met the entry criteria for that trial and completed A0081066 study through visit 7

Exclusion Criteria:

* Experienced serious adverse event during the A0081066 trial that was considered related or possibly related to study medication by the investigator or sponsor
* non-compliant during A0081066 trial
* clinically significant or unstable medical condition both HIV-related and non-HIV related including but not limited to, cardiac, pulmonary or hepatorenal disease that, in the opinion of the investigator, would compromise participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (27):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, West Hollywood, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Safety Harbor, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Seattle, Washington
- Puerto Rico (2):
  - Pfizer Investigational Site, Ponce
  - Pfizer Investigational Site, San Juan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081095&StudyName=Open%20Label%20Safety%20And%20Efficacy%20Study%20Of%20Pregabalin%20In%20Subjects%20With%20Nerve%20Pain%20Asociated%20With%20HIV%20Neuropathy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: With completion of A0081066 (NCT00232141), subjects had option of initiating treatment with pregabalin under open-label conditions for 3 months in A0081095, an open-label extension trial. Treatment in A0081095 was initiated on the evening of the subjects' Visit 7/Termination Visit in A0081066. A0081095 was conducted in the United States.
Groups:
- Pregabalin: Subjects who met all eligibility criteria initiated open-label treatment at 150 mg/day (75 mg BID). Further adjustments of total daily dose within the dose range 150 to 600 mg/day (BID) were permitted throughout the study to optimize pain control and minimize adverse events (AEs).
Period: Overall Study
Arm/Group | Pregabalin
Started | 220
Completed | 190
Not Completed | 30
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 11
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 178

OUTCOME MEASURES:

1. Primary Outcome: Mean Visual Analogue Scale (VAS) Pain Scores
Description: Pain scores were assessed on a 100 mm Visual Analogue Scale (VAS); scores range from 0= no pain to 100= worse pain. Subjects assessed their pain during the last week.
  Endpoint = last non-missing observation carried forward after Baseline visit.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Endpoint
Population: The full analysis set was defined as all subjects who met all eligibility criteria and took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 220
score on scale
  Baseline (n=203) | 38.61 (27.10)
  Week 4 (n=204) | 30.75 (25.19)
  Week 8 (n=200) | 30.16 (25.78)
  Week 12 (n=207) | 28.95 (26.05)
  Endpoint (n=217) | 29.39 (26.32)

ADVERSE EVENTS:
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 10
Other Adverse Events (participants affected / at risk) | 82
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pregabalin
Cellulitis (Infections and infestations) | 2/220
Pneumonia (Infections and infestations) | 1/220
Alcohol poisoning (Injury, poisoning and procedural complications) | 1/220
Chest pain (General disorders) | 1/220
Ankle fracture (Injury, poisoning and procedural complications) | 1/220
Syncope (Nervous system disorders) | 1/220
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/220
Abscess limb (Infections and infestations) | 1/220
Streptococcal infection (Infections and infestations) | 1/220
Pancreatitis (Gastrointestinal disorders) | 1/220
Deep vein thrombosis (Vascular disorders) | 1/220
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pregabalin
Dizziness (Nervous system disorders) | 22/220
Somnolence (Nervous system disorders) | 21/220
Peripheral edema (General disorders) | 13/220
Diarrhea (Gastrointestinal disorders) | 12/220
Fatigue (General disorders) | 11/220
Euphoric mood (Psychiatric disorders) | 8/220
Headache (Nervous system disorders) | 8/220
Cough (Respiratory, thoracic and mediastinal disorders) | 7/220
Dry mouth (Gastrointestinal disorders) | 7/220
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7/220
Vomiting (Gastrointestinal disorders) | 7/220
Nausea (Gastrointestinal disorders) | 6/220
Back pain (Musculoskeletal and connective tissue disorders) | 6/220
Upper respiratory tract infection (Infections and infestations) | 5/220
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5/220
Rash (Skin and subcutaneous tissue disorders) | 5/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.